CLINICAL TRIAL: NCT03933813
Title: Evaluation and Treatment of Iron Deficiency in Ovarian Cancer Patients Receiving Neoadjuvant Chemotherapy
Brief Title: Evaluation and Treatment of Iron Deficiency in Ovarian Cancer Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UW18106; 2019-0022 (Other: Institutional Review Board); A532820 (Other: UW Madison); SMPH/OB-GYN/GYN ONCOLOGY (Other: UW Madison); NCI-2019-02185 (Registry Identifier: NCI Trial ID); Protocol Version 8/15/2019 (Other: UW Madison)
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Epithelial Ovarian Cancer; Anemia; Iron Deficiency Anemia
Keywords: ovarian cancer; anemia; iron deficiency; blood transfusion
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Anemia; Anemia, Iron-Deficiency; Ovarian Neoplasms; Iron Deficiencies | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Intervention Model Description: Unblinded, window of opportunity trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IV Iron Sucrose (Experimental): Four intravenous iron sucrose infusions prior to debulking surgery administered as four 200mg infusions, given no less than 7 days apart over a 30 day +/- 7 day period
  Interventions: Other: Iron Sucrose

INTERVENTIONS:
Other: Iron Sucrose — Venofer (Iron Sucrose Injection USP) is a brown, sterile, aqueous, complex of polynuclear iron (III)-hydroxide in sucrose for intravenous use.
  Other Names: Venofer

SUMMARY:
This study tests the hypothesis that IV iron sucrose infusions given to iron deficient ovarian cancer patients prior to debulking surgery can improve pre-operative iron stores and decrease transfusion of packed red blood cells in the peri-operative period. 21 participants at least 18 years of age with epithelial ovarian cancer of any stage requiring neoadjuvant chemotherapy and surgery will be enrolled. Participants will be on study for a period of up to 3 months.

DETAILED DESCRIPTION:
Iron deficiency and anemia are common in cancer patients. Data from the University of Wisconsin (UW) suggest that more than 50% of ovarian cancer patients undergo blood transfusion during their cancer treatments. Transfusion rates are particularly high in patients who receive neoadjuvant chemotherapy (NACT), despite multiple opportunities to diagnose and treat anemia prior to surgery. Blood transfusions have been associated with worse survival in ovarian cancer patients. Seventy-seven percent of ovarian cancer patients who receive NACT at the UW are anemic prior to surgery, and the same percentage receive a perioperative blood transfusion, defined as a blood transfusion within 72 hours of surgery. Iron deficiency without anemia is also common in cancer patients, though little has been published regarding how frequently it occurs in ovarian cancer patients. Functional iron deficiency, a lack of iron incorporation into erythroid precursors despite adequate iron stores, is also common in cancer patients. Study investigators hypothesize that IV iron sucrose infusions given to iron deficient ovarian cancer patients prior to debulking surgery can improve pre-operative iron stores and decrease transfusion of packed red blood cells in the peri-operative period.

Eligible participants will have a new epithelial ovarian cancer diagnosis, with planned neoadjuvant chemotherapy and interval debulking surgery. The study cohort will consist of participants with iron deficiency without anemia (defined below) prior to starting chemotherapy. Iron deficient participants with anemia are already offered iron sucrose infusions as part of their standard of care treatment.

The study group will include participants with planned neoadjuvant chemotherapy and debulking surgery with a normal Hgb within 30 days of study enrollment. Iron studies including ferritin, transferrin, total iron binding capacity (TIBC), reticulocyte count and serum iron, will be performed on these participants for research purposes only. Consent will be obtained prior to drawing research-related iron studies. The majority of participants will have Hgb levels available in their records from the last 30 days, either from the UW, or from a referring institution. If this is not the case, pre-chemotherapy lab studies will be obtained the day of their visit, which would routinely include a Hgb level.

Participants will sign a consent to receive four IV iron sucrose transfusions, prior to their debulking surgery, and be followed for prospective data collection. Consent will be signed for the infusion and for prospective data collection related to future laboratory studies and rates of transfusion of blood products. Participants with a normal Hgb and normal iron studies will participate in the prospective data collection portion of this study only. Prospective data collection will continue until subjects have completed first-line chemotherapy.

Subjects will be enrolled until 21 evaluable participants have been enrolled. Evaluable participants will have true or functional iron deficiency without anemia and have received at least one IV iron sucrose infusion.

Iron studies will be repeated 21 days (+/- 7 days) after last infusion in participants who receive IV iron sucrose. Participants with persistent iron deficiency will be referred to hematology.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Has a diagnosis of true or functional iron deficiency without anemia within 30 days of treatment on this protocol

  * Iron deficiency without anemia (normal Hgb >/= 11.6 g/dL but ferritin < 30 ng/mL)
  * Functional iron deficiency without anemia (ferritin >30 ng/ml and iron saturation of <50%)
* Has a clinical diagnosis of suspected epithelial ovarian cancer based on imaging studies, exam findings and laboratory values
* Participants must be planning to receive neoadjuvant chemotherapy for their cancer diagnosis (NACT is defined as chemotherapy prior to debulking surgery)
* Participants must be planning to undergo surgery for their cancer diagnosis
* Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to administration of first dose of IV iron sucrose. WOCBP is defined as patients who retain their reproductive structures and are not menopausal (defined as > age 50 with no menses for at least 1 year)
* Participants of reproductive potential must agree to use effective birth control during study participation. Effective birth control is defined as any FDA approved contraceptive method

Exclusion Criteria:

* Currently taken any form of oral or intravenous iron therapy. Patients must have discontinued iron therapy > 30 days from study entry
* Current untreated or unstable heart disease
* History of iron induced hypersensitivity or allergy
* History of leukemia, lymphoma, or other myelodysplastic disorders
* Prior diagnosis of hemochromatosis or hemoglobinopathy (e.g. thalassemia)
* Any subject with immediate requirement for radiotherapy
* Concomitant enrollment in another clinical trial interfering with endpoints on this study
* Any medical condition which could compromise participation in the study according to the investigator's assessment
* Female patient who is pregnant or breast-feeding
* Patients unwilling or unable to comply with the protocol or unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Rate of Peri-operative Blood Transfusion | Within 72 hours of surgery, up to 5 weeks on study
  Defined as a transfusion of Packed Red Blood Cells (PRBCs) within 72 hours of surgery, in iron deficient ovarian cancer patients who receive IV iron sucrose therapy prior to surgery compared to a historical controls (historically 77%). The primary endpoint will be summarized with descriptive statistics and conducted using a Fisher's exact test and exact binomial confidence intervals. Point estimates and exact 95% confidence intervals (CI) will be calculated.

SECONDARY OUTCOMES:
Rate of Iron Deficiency Anemia | up to 21 days following surgery
  The rate of iron deficiency anemia in all ovarian cancers patients at the University of Wisconsin. This endpoint will be summarized with descriptive statistics and conducted using a Fisher's exact test and exact binomial confidence intervals. In particular, point estimates and exact 95% confidence intervals (CI) will be calculated.
Rate of Resolution of Iron Deficiency Anemia After Intervention | up to 21 days following surgery
  Iron deficiency anemia is defined as ferritin > 30 ng/mL and iron saturation of < 50%.
  This endpoint will be summarized with descriptive statistics and conducted using a Fisher's exact test and exact binomial confidence intervals. In particular, point estimates and exact 95% confidence intervals (CI) will be calculated.
Incidence of Treatment Emergent Adverse Events (AEs) | up to 21 days following surgery
  Safety and Tolerability will be monitored by measuring adverse events data with date of onset (or worsening) on or after the start-date treatment with iron sucrose and end of study (post-operative visit (7 to 21 days following surgery). AEs are defined as mild, moderate and severe.
  This endpoint will be summarized with descriptive statistics and conducted using a Fisher's exact test and exact binomial confidence intervals. In particular, point estimates and exact 95% confidence intervals (CI) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Barroilhet, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/